CLINICAL TRIAL: NCT03098836
Title: Prospective Study of Apalutamide and Abiraterone Acetate iN ChemoTHerapy-Naïve mEn With mCRPC Stratified by Race
Brief Title: Apalutamide and Abiraterone Acetate in African American and Caucasian Men With Metastatic Castrate Resistant Prostate Cancer
Acronym: PANTHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daniel George, MD (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Daniel George, MD, Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00075097
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: metastatic; castrate resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — apalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Caucasian (Experimental)
  Interventions: Drug: ARN-509; Drug: Abiraterone Acetate; Drug: Prednisone
- African American (Experimental)
  Interventions: Drug: ARN-509; Drug: Abiraterone Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: ARN-509 — 240 mg orally daily
  Other Names: apalutamide
Drug: Abiraterone Acetate — 1000 mg orally daily
  Other Names: Zytiga
Drug: Prednisone — 5 mg orally twice daily (for total daily dose 10 mg)

SUMMARY:
The primary goal is to prospectively estimate the median PFS of African American and Caucasian men with mCRPC taking apalutamide, abiraterone acetate, and prednisone. Secondary objectives include: PSA kinetics: to determine the duration of PSA response, time to nadir, and percent of men who achieve a PSA < 0.1; Radiographic assessments: to estimate the rate of objective response and incidence of bone flares; Safety (NCI CTC v4.0) and tolerability, particularly incidence and grade of hypertension in the two populations.

This is a non-comparative pilot open-label, parallel arm, multicenter study of apalutamide and abiraterone acetate in African American and Caucasian men with mCRPC. It is anticipated that 3 additional sites will be needed to accrue 100 subjects (50 African American and 50 Caucasian) over a 24 month accrual period. The study agents will be administerd at the following doses: apalutamide 240mg orally once daily, abiraterone acetate 1000mg orally once daily, and prednisone 5 mg BID in 4-week cycles throughout the treatment period.

Fifty (50) patients will be enrolled in each group (AA and Caucasians). The proportion of patients who experience PSA decline of 30%, 50% and 90% will be estimated with exact 95% confidence intervals based on the binomial distribution will be computed. In addition, post therapy changes in PSA will be explored as a continuous outcome. The Kaplan-Meier product limit method will be used to estimate the rPFS, biochemical PFS and overall survival distributions.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age ≥ 18 years
2. Karnofsky performance status ≥ 70 (Appendix 1)
3. Life expectancy of ≥ 12 months as determined by treating investigator
4. Written Authorization for Use and Release of Health and Research Study Information (HIPAA authorization per institutional requirements)
5. Willing/able to adhere to the prohibitions and restrictions specified in this protocol
6. Willing to take abiraterone acetate on an empty stomach, and should be able to swallow tablets whole, without crushing/chewing tablets. Must have the ability to swallow, retain, and absorb oral medication.
7. Medications known to lower the seizure threshold (see list under prohibited meds, appendix 2) must be discontinued or substituted at least 4 weeks prior to study entry
8. Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug. Abstinence is an acceptable method of birth control.
9. Adequate bone marrow function as shown by: ANC ≥ 1.0 x 109/L, Platelets ≥ 100 x 109/L, Hb≥9 g/dL, (independent of transfusion and/or growth factors within 3 months prior to Cycle 1 Day 1)
10. Serum potassium ≥ 3.5 mEq/L
11. Serum albumin of ≥ 3.0 g/dl
12. AST/SGOT and ALT/SGPT <2.5 x Institutional Upper Limit of Normal (ULN)
13. Serum total bilirubin ≤ 1.5 x Institutional ULN (Note: In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, subject may be eligible)
14. GFR ≥45 mL/min
15. Histologically confirmed diagnosis of adenocarcinoma of the prostate. Histologic variants of prostate cancer comprising of >50% of the tumor including neuroendocrine features and small cell carcinoma of the prostate are excluded.
16. Radiographic evidence of metastatic disease based on RECIST 1.1 Criteria OR by prostate cancer-specific PET imaging. Evaluable non-target lesions and/or bone only metastasis are permitted per RECIST 1.1 and PCWG3 guidelines. Non-target, pathological lymph nodes ≥ 10 mm and less than 15 mm in the short axis are permitted.
17. Ongoing ADT using an LHRH agonist (e.g. leuprolide, goserelin) or antagonist (e.g. degarelix) must continue on therapy unless prior bilateral orchiectomy has been performed.
18. PSA ≥ 2.0 ng/mL
19. Evidence of castration resistant disease in the setting of ongoing ADT (medical or surgical) as evidenced by one of the following:

    * Absolute rise in PSA of 2.0 ng/mL or an increase >25% from the nadir, minimum 2 consecutive rising PSA levels with an interval of ≥ 1 week between each PSA level, OR
    * CT or MRI based evidence of disease progression (soft tissue, nodal or visceral disease progression) according to PCWG3 criteria or RECIST 1.1 criteria, OR
    * At least 1 new bone scan lesion as compared to the most immediate prior radiologic studies.
20. A minimum of 2 weeks elapsed off of antiandrogen therapy prior to start of study drug (i.e. flutamide, nilutamide, bicalutamide.)
21. A minimum of 2 weeks elapsed off of sipuleucel-T and radiation therapy prior to start of study drug
22. A minimum of 4 weeks from any major surgery prior to start of study drug.
23. Self-reported race of either African American or Caucasian.
24. Ability to understand and the willingness to sign a written informed consent document. If the subject is unable to understand the consent due to comorbidity, such as Alzheimer's disease, consent by a legally authorized representative and assent by the subject will be obtained.

Exclusion Criteria:

1. Prior treatment with abiraterone acetate, enzalutamide, apalutamide (ARN-509), galaterone (TOK-001), orteronel (TAK-700), or similar agent
2. Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
3. Active or symptomatic infection including HIV, viral hepatitis or chronic liver disease
4. Any chronic medical condition requiring a higher dose of corticosteroid than 5mg prednisone/prednisolone bid
5. Have known allergies, hypersensitivity, or intolerance to abiraterone acetate, apalutamide or prednisone or their excipients.
6. Pathological finding consistent with small cell carcinoma of the prostate
7. Symptomatic liver or visceral organ metastasis
8. Have a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
9. Known brain metastasis
10. Prior cytotoxic chemotherapy or biologic therapy for the treatment of CRPC. Note: sipulecel-T is permitted with a 2-week washout.
11. Previously treated with ketoconazole for prostate cancer for greater than 7 days
12. Prior systemic treatment with an azole anti-fungal drug (e.g. fluconazole, itraconazole) within 4 weeks of Cycle 1, Day 1.
13. Uncontrolled hypertension (systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg). Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
14. Poorly controlled diabetes, FBS ≥200 mg/dL
15. History of pituitary or adrenal dysfunction
16. Symptomatic Atrial Fibrillation, or other symptomatic cardiac arrhythmia
17. Other malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of recurrence within 24 months
18. History of any of the following:

    * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 6 months of Cycle 1 Day 1, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy)
    * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to first dose of study drug. Venous thrombolic events within 6 months are permitted IF they are not attributed to prostate cancer (in the opinion of the treating physician).
19. Avoid concomitant strong CYP3A4 inducers during abiraterone acetate treatment.
20. Avoid co-administration of abiraterone acetate with CYP2D6 substrates that have a narrow therapeutic index. If an alternative treatment cannot be used, exercise caution and consider a dose reduction of the concomitant CYP2D6 substrate
21. Baseline moderate or severe hepatic impairment (Child Pugh Class B & C)
22. Use of herbal products that may decrease PSA levels (i.e., saw palmetto) refer to section 8.3.2 (no washout period required)
23. Administration of an investigational therapeutic within 30 days prior to Cycle 1, Day 1
24. Any condition which, in the opinion of the investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. George, MD, Principal Investigator — Duke Cancer Institute
Locations (14):
- United States (14):
  - Tulane University, New Orleans, Louisiana
  - Chesapeake Urology Associates, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Cancer Center, Chapel Hill, North Carolina
  - Johnston Hematology and Oncology of Clayton, Clayton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Scotland Memorial Hospital, Laurinburg, North Carolina
  - Southeastern Regional, Lumberton, North Carolina
  - Johnston Memorial Hospital, Smithfield, North Carolina
  - Spartanburg Regional, Spartanburg, South Carolina
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Caucasian: Self-identified Caucasian patients with mCRPC
- African American: Self-identified African American patients with mCRPC
Period: Overall Study
Arm/Group | Caucasian | African American
Started | 50 | 43
Completed | 14 | 22
Not Completed | 36 | 21
Not completed — Adverse Event | 1 | 3
Not completed — Lack of Efficacy | 30 | 15
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caucasian | African American | Total
Number analyzed (Participants) | 50 | 43 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (7) | 70 (9) | 70 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 43 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 43 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 43 | 43
  White | 50 | 0 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 43 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 2-Year Progression-Free Survival (PFS)
Description: Radiographic PFS based on PCWG2 criteria or based on the onset of a skeletal related event. Imaging obtained every 12 weeks. Kaplan-Meier estimate of percentage of participants is reported.
Time Frame: every 12 weeks, up to 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Caucasian | African American
Number analyzed (Participants) | 50 | 43
Percentage of participants | 38 [27 to 55] | 61 [48 to 78]

2. Secondary Outcome: 2-year PSA Progression Free Survival
Description: PSA progression-free survival
Time Frame: every 4 weeks, up to 2 years
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Caucasian | African American
Number analyzed (Participants) | 50 | 43
percent | 38 [24 to 58] | 60 [46 to 80]

3. Secondary Outcome: Time to PSA Nadir
Description: Time to PSA nadir
Time Frame: every 4 weeks, up to 2 years
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- African American: Self-identified Caucasian patients with mCRPC
Arm/Group | Caucasian | African American
Number analyzed (Participants) | 50 | 43
months | 1.9 [1.0 to 5.5] | 5.3 [1.8 to 8.3]

4. Secondary Outcome: Percent of Men Who Achieve a PSA < 0.1
Description: Percent of men who achieve a PSA < 0.1
Time Frame: every 4 weeks, up to 2 years
Measure: Number; unit: percent of participant
Arm/Group | Caucasian | African American
Number analyzed (Participants) | 50 | 43
percent of participant | 26 | 40

5. Secondary Outcome: Radiologic Response Rates
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions assessed by CT: Complete Response (CR), disappearance of all lesions and any pathologic lymph nodes (target or non-target) must have reduction in short axis to <10 mm; Partial Response (PR), ≥30% decrease in the sum diameter of target lesions as compared to the baseline sum diameter; Overall Response (OR) = CR + PR
Time Frame: every 12 weeks, up to 2 years
Population: Four patients were unevaluable. Two patients did not have response recorded.
Measure: Number; unit: percent
Arm/Group | Caucasian | African American
Number analyzed (Participants) | 46 | 41
percent | 10 | 14

6. Secondary Outcome: Percentage of Participants With Bone Flares
Description: Percentage of participants who experienced bone flares per radiographic assessments
Time Frame: 12 weeks
Measure: Number; unit: percent
Arm/Group | Caucasian | African American
Number analyzed (Participants) | 50 | 43
percent | 16 | 9

7. Secondary Outcome: Percentage of Participants With Hypertension
Description: Safety (NCI CTC v4.0) and tolerability, particularly incidence and grade of hypertension in the two populations. Grade assessed according to NCI CTC v4.0 with higher grade being worse is reported.
Time Frame: up to 2 years
Measure: Number; unit: percent of participants
Arm/Group | Caucasian | African American
Number analyzed (Participants) | 50 | 43
percent of participants
  Grade 2 hypertension | 40 | 40
  Grade 3 hypertension | 16 | 14
  Grade 4 hypertension | 0 | 2

8. Secondary Outcome: Median Overall Survival
Description: Survival of subjects over the time the study is ongoing
Time Frame: every 6 months, up to 82 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Caucasian | African American
Number analyzed (Participants) | 50 | 43
months | 36 [30 to 60] | 72 [44 to NA] — Upper confidence interval limit not estimable due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: up to 2 years, while participant was receiving study drugs; all-cause mortality was collected throughout the follow-up period (up to 82 months)
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.4.0.
Arm/Group | Caucasian | African American
All-Cause Mortality (participants affected / at risk) | 34/50 | 20/43
Serious Adverse Events (participants affected / at risk) | 12/50 | 10/43
Other Adverse Events (participants affected / at risk) | 50/50 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caucasian (N=50) | African American (N=43)
Coronary Artery Blockage x4 (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Encephalitis infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3
CLOSED FRACTURE, HEAD (Injury, poisoning and procedural complications) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Study Drug Overdose (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
RHABDOMYOLSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
metastatic castration-resistant prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 1
Multifocal Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LAPAROSCOPIC COLECTOMY FOR COLON CANCER (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caucasian (N=50) | African American (N=43)
Anemia (Blood and lymphatic system disorders) | 5 | 7
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 3 | 5
Hyperthyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 4 | 3
Dry eye (Eye disorders) | 1 | 0
DANDRUFF (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Floaters (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 8
Diarrhea (Gastrointestinal disorders) | 11 | 8
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Dysphagia (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 10
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 7
Colitis (Gastrointestinal disorders) | 0 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Edema limbs (General disorders) | 3 | 4
Fatigue (General disorders) | 27 | 19
Fever (General disorders) | 1 | 0
Gait disturbance (General disorders) | 3 | 3
Irritability (General disorders) | 1 | 0
Localized edema (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 3
Pain (General disorders) | 10 | 9
Chills (General disorders) | 0 | 1
Edema face (General disorders) | 0 | 3
Facial pain (General disorders) | 0 | 1
Flu like symptoms (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 2
Bronchial infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 2
Rash pustular (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 4
Lung infection (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 5 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 4
Fracture (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3
Alkaline phosphatase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood bilirubin increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 1 | 7
Platelet count decreased (Investigations) | 4 | 1
Weight loss (Investigations) | 3 | 8
White blood cell decreased (Investigations) | 3 | 4
Creatinine increased (Investigations) | 0 | 2
Weight gain (Investigations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalemia (Metabolism and nutrition disorders) | 15 | 23
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 13
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Cognitive disturbance (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Concentration impairment (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Dizziness (Pregnancy, puerperium and perinatal conditions) | 5 | 6
Dysarthria (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Dysgeusia (Pregnancy, puerperium and perinatal conditions) | 7 | 4
Headache (Pregnancy, puerperium and perinatal conditions) | 6 | 7
Intracranial hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Memory impairment (Pregnancy, puerperium and perinatal conditions) | 2 | 3
Paresthesia (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Presyncope (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Seizure (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Somnolence (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Spasticity (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Tremor (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Extrapyramidal disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Neuralgia (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Peripheral sensory neuropathy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Syncope (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Transient ischemic attacks (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 4 | 0
Confusion (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 7 | 4
Hallucinations (Psychiatric disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 4 | 1
Renal calculi (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 6 | 5
Urinary incontinence (Renal and urinary disorders) | 5 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 3
Gynecomastia (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 5
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 8 | 3
Hypertension (Vascular disorders) | 28 | 24
Hypotension (Vascular disorders) | 1 | 2
Thromboembolic event (Vascular disorders) | 1 | 2
PULMONARY ARTERY EMBOLISM, CT CHEST FINDINGS (Vascular disorders) | 1 | 0
PREMATURE VENTRICULAR CONTRACTIONS (Cardiac disorders) | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
ELEVATED HEART RATE (Cardiac disorders) | 1 | 0
EXCESSIVE SALIVA (Gastrointestinal disorders) | 0 | 1
CANKER SORES IN MOUTH (Gastrointestinal disorders) | 1 | 0
TONGUE ULCERS (Gastrointestinal disorders) | 1 | 0
MILD DIVERTICULITIS OF DESCENDING COLON AND SIGMOID COLON (Gastrointestinal disorders) | 1 | 0
PAIN, SHOULDERS (General disorders) | 1 | 0
MEDICATION OVERDOSE (General disorders) | 0 | 3
ACCIDENTAL OVERDOSE (General disorders) | 0 | 1
EDEMA (General disorders) | 0 | 1
HAIR LOSS (General disorders) | 0 | 1
HEAD PAIN (General disorders) | 1 | 0
POSTERIOR BILATERAL PELVIC ACHES (General disorders) | 1 | 0
VIVID DREAMS (Nervous system disorders) | 2 | 0
FEELING "WIRED" (Nervous system disorders) | 0 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0
COLD LIKE SYMPTOMS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAMMER TOE CORRECTION (Surgical and medical procedures) | 0 | 1
SKIN BIOPSIES (Surgical and medical procedures) | 1 | 0
LYMPH NODE BIOPSY (Surgical and medical procedures) | 0 | 1
MOH'S PROCEDURE ON NOSE (Surgical and medical procedures) | 1 | 0
LEFT HIP ARTHROPLASTY (Surgical and medical procedures) | 0 | 1
L - EXTRACTION CATARACT EXTRACAPSULAR WITH PHACO WITH INSERTION INTRAOCULAR PROSTHESIS (Surgical and medical procedures) | 0 | 1
RIGHT INTERNAL CAROTID ARTERY STENT (Surgical and medical procedures) | 1 | 0
PROVENGE INFUSION (Surgical and medical procedures) | 0 | 1
CYSTOURETHROSCOPY, WITH INSERTION OF INDWELLING STENT, UROGRAPHY RETROGRADE (Surgical and medical procedures) | 0 | 1
MOHS SURGERY (Surgical and medical procedures) | 1 | 0
TRANSIENT HYPERTENSION INCREASE RELATED TO BENADRYL (Vascular disorders) | 0 | 1
NONSUSTAINED VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0
ERYTHEMA OF FACE; OCCURS WITH FEVER (Infections and infestations) | 1 | 0
NON FASTING GLUCOSE ELEVATED (Investigations) | 0 | 1
HYPERLIPIDEMIA (Investigations) | 1 | 0
URINE ODOR (Renal and urinary disorders) | 1 | 0
STRONG URINE ODOR (Renal and urinary disorders) | 1 | 0
MALODOROUS URINE (Renal and urinary disorders) | 0 | 1
URINARY HESITANCY (Renal and urinary disorders) | 0 | 1
URETER SPASM (Renal and urinary disorders) | 0 | 2
INTERMITTENT BURNING WITH URINATION (Renal and urinary disorders) | 0 | 1
INTERMITTENT SULFUR SMELL AFTER TAKING APALUTAMIDE (Renal and urinary disorders) | 0 | 1
NOCTURIA (Renal and urinary disorders) | 1 | 0
INGROWN TOENAIL (Skin and subcutaneous tissue disorders) | 0 | 1
BOILS (Skin and subcutaneous tissue disorders) | 1 | 0
NASAL SORES (Skin and subcutaneous tissue disorders) | 1 | 0
NAIL THINNING (Skin and subcutaneous tissue disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
PIMPLE ON SCROTUM (Skin and subcutaneous tissue disorders) | 0 | 1
BUMP ON R AND L BUTTOCKS (Skin and subcutaneous tissue disorders) | 0 | 1
DARK UNDER EYE CIRCLES (Skin and subcutaneous tissue disorders) | 1 | 0
CHILL ON BACK AND LEGS (Skin and subcutaneous tissue disorders) | 0 | 1
RASH, RIGHT WRIST AND UPPER ARM (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN LESION CAUTERIZATION (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATOSIS PAPULOSANIGRA (Skin and subcutaneous tissue disorders) | 0 | 1
LEFT FOREARM LACERATION (Skin and subcutaneous tissue disorders) | 0 | 1
BILATERAL FOOT CALLOUS (Skin and subcutaneous tissue disorders) | 0 | 1
DISCOLORED HANDS (Skin and subcutaneous tissue disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 2
INT NIGHT SWEATS (Endocrine disorders) | 0 | 1
ELEVATED TSH (Endocrine disorders) | 1 | 1
ELEVATED CREATININE (Renal and urinary disorders) | 0 | 1
RASH RIGHT WRIST AND UPPER ARM (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITIC HYPERPIGMENTED LESION ON BACK (Skin and subcutaneous tissue disorders) | 0 | 1
DISCOLORATION IN HANDS (Skin and subcutaneous tissue disorders) | 0 | 1
RASH ON TORSO (Skin and subcutaneous tissue disorders) | 1 | 0
HAIR LOSS ON CHEST (Skin and subcutaneous tissue disorders) | 1 | 0
LEFT KNEE NUMBNESS (General disorders) | 0 | 1
LEFT BIG TOE TENDERNESS (General disorders) | 0 | 1
TSH ELEVATED (Investigations) | 2 | 0
COVID (Investigations) | 0 | 1
PSA INCREASED (8.41) (Investigations) | 1 | 0
PULLED GROIN MUSCLE (Musculoskeletal and connective tissue disorders) | 1 | 0
CRAMPING IN HANDS (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERMITTENT BILATERAL HAND AND FOOT CRAMPS (Musculoskeletal and connective tissue disorders) | 1 | 0
LEFT JAW CLICKING (Musculoskeletal and connective tissue disorders) | 0 | 1
SHOULDER TENDERNESS L (Musculoskeletal and connective tissue disorders) | 0 | 1
CHEST CONGESTION (Musculoskeletal and connective tissue disorders) | 1 | 0
LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1 | 0
RESTLESS LEG SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0
RIGHT HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT03098836/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03098836/SAP_001.pdf